CLINICAL TRIAL: NCT03162523
Title: Norwegian Experiences With Interstitial Radiation Treatment (Brachytherapy) for Men With High-risk Localised Prostate Cancer
Brief Title: Experiences With HDR-brachytherapy in Norway
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Principal Investigator, Trude Baastad Wedde, Consultant oncologist, Oslo University Hospital
Other Study IDs: 677905
Record Dates: First submitted 2017-05-07; First posted 2017-05-22 (Actual); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Scandinavian Prostate Cancer Group (SPCG), study number 7: Patients included in hallmark study of SPCG-7 receiving EBRT to 70 Gy in combination with lifelong anti-androgen treatment
  Interventions: Radiation: High-Dose Rate Brachytherapy
- Norwegian Urologic Cancer Group (NUCG) study number 7: Patients receiving EBRT to 74 Gy in combination with hormonal therapy. Approved by ethical comittee. Questionnaires already been completed during a different study (NUCG-7). These patients will therefore not be contacted again.
  Interventions: Radiation: High-Dose Rate Brachytherapy

INTERVENTIONS:
Radiation: High-Dose Rate Brachytherapy

SUMMARY:
There are 3 articles that will be written about the experience with HDR-brachytherapy (HDR-BT) in patients with high-risk prostate cancer in Norway as part of a doctorial thesis-project. The project will focus on survival, side-effects and dosimetry variables as the main points of interest.

DETAILED DESCRIPTION:
First article will compare overall and prostate cancer specific-mortality in patients who has received HDR-BT compared to patients who has received external beam radiation therapy only (EBRT). Patients who have been treated with HDR-BT have been enrolled in an approved registry at Oslo University Hospital since 2004. The control group (EBRT only) data are from the Lancet published hallmark study SPCG-7 (Scandinavian Prostate Cancer Group). This is a case-control study.

Second article will focus on side-effects of HDR-BT compared to EBRT patients. Patients included in the registry described above have been sent (and completed with a 72% answer rate) a questionnaire of the standard Expanded Prostate Cancer Index (EPIC-26) form. This will be compared to patients who already have answered the same questionnaire in a previously published study (approved by the Norwegian Ethical Committee).

The Third article will investigate if there are any association between patients reporting severe adverse effects after HDR-BT and the patients dosimetry reports (i.e are there a larger dose to the urethra or rectum in these patients?)

ELIGIBILITY:
Inclusion Criteria:

* age, high-risk prostate cancer, general good Health, anatomical favourable condition for brachytherapy

Exclusion Criteria:

* poor Health, metastasis, T3b stage tumour, Prostate Specific Antigen (PSA) Levels > 75, biological age > 75 years

Max Age: 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Men are included from the south-east area of Norway and for control Groups from the entire country so that the study population is generalised.
Sampling Method: Non-Probability Sample
Enrollment: 325 (Actual)
Dates: Start 2004-01 (Actual); Primary Completion 2016-10-15 (Actual); Study Completion 2016-10-15 (Actual)

PRIMARY OUTCOMES:
Overall- and Prostate-Cancer specific mortality in patients treated with HDR-BT compared to EBRT alone | 24 weeks
  The final measured outcome is death by prostate cancer, death due to other cause (overall mortality) or alive at 10 years.
Patient-reported side-effects after HDR-BT compared to conventional EBRT | 1 year
  Patient self-reported side-effects focusing on rectal, bladder, quality of life, sexual function and psycological bother will be recorded in both Groups and compared.
Are there an Association between rectal dosage after HDR-BT and self-reported rectal bother in patients undergone HDR-BT treatment ? | 2 years
  Investigations into needle placement, dosage and anatomical variations will be examined in patients who report rectal problems 5 years after HDR-BT treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Trude Wedde, MD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No